CLINICAL TRIAL: NCT07356817
Title: Cardiovascular Risk Assessment in Young Women After Index Pregnancy With and Without Placental Complications
Acronym: CARDIOMOM
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Hospital Sant Joan de Deu (Other); Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-MOM-2022-87
Record Dates: First submitted 2025-11-14; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular (CV) Risk; Preeclampsia (PE); Fetal Weight
Keywords: preeclampsia; Cardiovascular Risk; app
MeSH Terms: conditions — Pre-Eclampsia; Fetal Weight; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood, urine and hair samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young women with an index pregnancy with and without placental complications: CV biophysical, imaging and biochemical variables 3-6 years after index pregnancy (approximate n=1260) will be evaluated. Analyses will include urbanome, placental function and perinatal variables during index pregnancy and postnatal variables such as maternal socio-economic status, lifestyle, urban exposome, mental health, blood pressure, cardiac function, coronary artery disease by Coronary Computed Tomography (CCT) and CCT angiography, RM Quantitative Myocardial Perfusion, ophthalmic artery index, carotid intima- media thickness up to 6 years after delivery to predict higher risk for CVD later in life. Patients' needs and expectations according to CV health would be evaluated.

SUMMARY:
In this project, the investigators aim to study how all these factors determine the cardiovascular status of a total of 1,800 mothers, 3 to 6 years after delivery. In addition, the investigators want to assess whether lifestyle and living conditions after childbirth may improve or worsen this imprint, since women often prioritize their families over themselves, making it more difficult to maintain a healthy lifestyle that could reduce their cardiovascular risk. Furthermore, the investigators will evaluate how environmental exposures influence their health, as well as explore potential strategies for prediction and prevention.

The goal is to develop an easy-to-use algorithm or test that allows women and their physicians to assess this risk, ideally in the form of a mobile app. Although predictive algorithms for cardiovascular health already exist, most have been developed using predominantly male or older populations, and none have taken into account pregnancy-related events or environmental exposure - both of which are key determinants of women's cardiovascular health.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the leading cause of death among women, particularly non-obstructive myocardial infarction, heart failure, and stroke. However, neither women themselves nor, often, their physicians are fully aware of this reality. This lack of awareness is partly due to gender-related myths and biases that have led to insufficient study of the specific causes and risk factors that affect women's cardiovascular systems. Traditionally, it has been assumed that cardiovascular risk mechanisms, prediction, diagnosis, and treatment are the same in men and women. Today, it is known that this is not true: while the severity and mortality due to cardiovascular disease have decreased in men, they continue to rise and remain more severe among women.

Reproductive history and hormonal influence play a decisive role in modulating cardiovascular risk in women. Experiencing complications during pregnancy - such as preeclampsia (a hypertensive disorder caused by abnormal placental function), preterm delivery, or the birth of a low-weight infant - increases the risk of cardiovascular complications up to sevenfold later in life, compared with women who had normal pregnancies. This is explained by the fact that the cardiovascular system undergoes major adaptive changes during pregnancy; in complicated pregnancies, these adaptations fail to occur properly, resulting in cardiovascular stress and damage.

Among the objectives of this project, the investigators also aim to evaluate other risk factors such as lifestyle and external influences like exposure to environmental pollutants, which may further contribute to cardiovascular vulnerability. Pregnancy represents a critical window of susceptibility - as seen in other conditions such as COVID-19 - during which these environmental and biological impacts on the cardiovascular system are amplified.

In this project, the aim is to investigate how all these factors determine cardiovascular health in a cohort of 1,800 mothers, assessed 3 to 6 years after childbirth. The investigators will also examine how postnatal lifestyle and self-care behaviors may either mitigate or exacerbate this imprint. Women often prioritize their families' needs over their own, which can make it difficult to maintain healthy habits that reduce cardiovascular risk. Moreover, the investigators will study how environmental exposures influence maternal health and explore potential predictive and preventive strategies.

The goal is to develop an easy-to-use algorithm or test - ideally in the form of a mobile application - to help women and their physicians assess cardiovascular risk. Although predictive algorithms for cardiovascular health already exist, they have mostly been developed in predominantly male or older populations, and none have considered pregnancy-related factors or environmental exposures, both of which are key determinants of women's cardiovascular health.

To date, preventive cardiovascular strategies have not been specifically designed for women, and even less so for recently postpartum women. Existing tools have not been adapted for this population. This project brings together obstetricians and cardiologists, as well as midwives and primary care physicians - the healthcare professionals primarily responsible for women's health and well-being. The investigators believe that this multidisciplinary approach is crucial to anticipate cardiovascular disease and implement truly preventive strategies.

All study findings will be disseminated through educational sessions for healthcare professionals, new clinical tools and practices to improve patient satisfaction, audiovisual materials for better maternal health communication, and through professional societies (such as SEGO, SEC, SEAP, SEM, etc.). Results will also be published in open-access scientific journals and shared via public outreach, including media coverage, conferences in hospitals and community centers, social media (@DonaSantPau), and the institutional website (http://www.santpau.cat/web/public/go-inici

).

The active participation of women in this study will also allow the creation of discussion and advocacy groups among participants, supporting dissemination through social media, online platforms (https://inatal.org), and patient associations (such as El parto es nuestro), as well as newspapers, radio, and television.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in the BiSC (Barcelona Life Study Cohort), EuroPE (Randomized open-label control trial to evaluate if the incorporation of sFlt1/PlGF ratio in the diagnosis and classification of PE improves maternal and perinatal outcomes in women with suspicion of the disease; PI16/00375) and AngioCor (Cardiac dysfunction and remodeling in patients with preeclampsia regulated by antiangiogenic environment: clinical and experimental approach, PI19/00702) cohort studies
* Who have delivered within the previous 3-6 years.
* Give written consent when invited to participate in this study protocol.

Exclusion Criteria:

* Unwillingness to participate in this study
* Probability of loss to follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young women who presented an index pregnancy with and without placental complications, who have previously participated in cohort studies performed by our group identifying biophysical, biochemical, psychosocial and environmental cardiovascular risk factors during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 1260 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hypertension | 3-6 years after index pregnancy
  Presence of hypertension, defined as stage 1 hypertension (SBP of 130-139 or DBP of 80-89 mmHg)
Abnormal cardiac function | 3-6 years after index pregnancy
  Abnormal cardiac function in the echocardiographic ultrasound assessment. Abnormal values of the different parameters will be considered according to reference limits published in 2020 by the British Society of Echocardiography
Biochemical cardiac markers | 3-6 years after index pregnancy
  Abnormal biochemical cardiac markers: NTproBNP >300 ng/L or high-sensitivity troponin>30 ng/L
Coronary artery disease | 3-6 years after index pregnancy
  Signs of coronary artery disease by computer tomography (CCT) myocardial perfusion imaging (mild (CACS≥10 AU and <100 AU); moderate (CACS≥100 AU and <400 AU) and severe (CACS ≥400 AU)
Other cardiovascular major events | 3-6 years after index pregnancy
  Cardiovascular major events (ictus, coronary artery disease, cardiac insufficiency or myocardiopathy)

SECONDARY OUTCOMES:
Age | 3-6 years after index pregnancy
  Patient age
Pregnancy complications | 3-6 years after index pregnancy
  Preeclampsia, pregnancy complications, presence of fetal distress, perinatal mortality, neonatal morbidity, and neonatal mortality.
Antrophometric measurements | 3-6 years after index pregnancy
  Percentages of body fat, muscle mass, visceral fat
Blood pressure | 3-6 years after index pregnancy
  Systolic and Dyastolic blood pressure
Computer tomography (CCT) myocardial perfusion imaging and RM Quantitative Myocardial Perfusion | 3-6 years after index pregnancy
  Allows an accurate and reliable assessment of both coronary epicardial stenosis and myocardial CT perfusion imaging at rest and during pharmacologic stress in the same examination. CCT will be performed with a 256-slice CT scanner (Philips Healthcare scanner) with prospective ECG-triggering as previously described. First, a noncontrast CCT will be performed to calculate the CACS using the Agatston scoring method. Second, CCTA will be performed following sublingual nitroglycerin and injection of nonionic contrast (Iopromide, Ultravist, Bayer Healthcare, Berlin, Germany). The presence of any coronary plaque (noncalcified, calcified, or mixed) and the presence of significant stenosis (≥50%) was assessed in all 17 coronary segments. One of 2 assigned and experienced cardiovascular radiologists assessed the CT scans for each participant.
Cardiovascular markers in maternal blood | 3-6 years after index pregnancy
  Venous blood samples will be collected without anticoagulant to obtain serum. Troponin T and NTproBNP will be measured in ng/ml using automated electrochemiluminescence immunoassays on the Roche Cobas platform (Roche Diagnostics GmbH, Mannheim, Germany).Intra-and interassay coefficients of variation were found to be <5%.
Laboratory data measured in mg/dl | 3-6 years after index pregnancy
  glucose, uric acid, creatinine, VLDL, LDL, HDL, total cholesterol, triglycerides
Cardiovascular assessment according to IBERLIFERISK score | 3-6 years after index pregnancy
  A score >50% is considered as a high-risk for CVD.
Hair sampling for cortisol determination | 3-6 years after index pregnancy
  Hair samples will be cut with scissors from the region of the posterior vertex, as close to the scalp as possible. Considering that hair grows approximately 1 cm per month, 3 cm will be obtained in order to evaluate hair cortisol levels representative of the last 3 months. Samples will be stored (in a dark container at room temperature) until analysis by liquid chromatography mass spectrometry.
Diet and nutrition | 3-6 years after index pregnancy
  evaluated by means of the Short Diet Quality Screener by REGICOR (registre Gironí del Cor) and by means of the validated 14-item questionnaire of adherence to the Mediterranean diet. Escale from 1-31. The highest the score, the highest the adherence to the mediterranean diet.
Physical activity | 3-6 years after index pregnancy
  evaluated by means of the Physical Activity Questionnaire by REGICOR, a validated questionnaire for quantifying physical activity in our population. The short questionnaire estimates energy expenditure in total PA and by intensity (light, moderate, vigorous), and includes 2 questions about sedentary behavior and a question about occupational PA.
Stress | 3-6 years after index pregnancy
  evaluated by the Perceived Stress Scale (PSS) Questionnaire, validated for quantifying perceived stress in our population. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived this: Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Mental health | 3-6 years after index pregnancy
  evaluated by the Psychiatric Diagnostic Screening Questionnaire (PDSQ), a brief, psychometrically strong, self-report scale designed to screen for the most common disorders encountered in outpatient mental health settings and validated in our population. The final version of the questionnaire contains 13 subscales (major depressive disorder [MDD], bulimia, post-traumatic stress disorder [PTSD], panic disorder, agoraphobia, social phobia, generalized anxiety disorder [GAD], obsessive-compulsive disorder [OCD], alcohol abuse/dependence, drug abuse/dependence, somatization, hypochondriasis, and psychosis). Additionally, there is a six-item psychosis screen.
Smoking habit | 3-6 years after index pregnancy
  evaluated by the Fagerström Questionnaire, validated questionnaire for quantifying dependence on smoking in our population.
Women experiences and eHealth | 3-6 years after index pregnancy
  For this aim, a team of anthropologists with a long experience in the fields of health and reproduction will use qualitative methods to understand the needs of women with and without CV risk after pregnancy. To this end, semistructured interviews will be undertaken with patients with low and high risk of CV disease. These interviews will be useful to have a deep understanding of the difficulties, desires, and needs in relation to interactions with practitioners and available services in healthcare settings. For proactive monitoring and follow-up of patients, a technological platform or App (CardioPlan), currently used for cardiac rehabilitation, will be restructured, which has a highly secure data repository located on the provider's server and then validated in a subgroup of patients (n=100).
BMI | 3-6 years after index pregnancy
  Weight and height will be combined to report BMI in kg/m^2
Waist/Hip ratio | 3-6 years after index pregnancy
  Measurements in cm2 of waist and hip to calculate waist/hip ratio in cm2
Heart rate | 3-6 years after index pregnancy
  Measured in hpm
Echocardiographic assesment | 3-6 years after index pregnancy
  Performed by a cardiologist specialized in cardiac imaging according to the usual standard protocol. High-resolution images will be acquired and post-processed with dedicated software for the speckle tracking analysis.
Myocardial deformation (strain) | 3-6 years after index pregnancy
  measured by echocardiography is increasingly recognized as a more effective technique than conventional ejection fraction (EF) in detecting subtle changes in left ventricular (LV) function and in predicting outcomes. AutoStrain TOMTEC Philips EPIQ CVx ultrasound systemwould be used for the analysis.
Carotid intima-media thickness | 3-6 years after index pregnancy
  Transverse longitudinal evaluation of the common carotid artery, its bifurcation and internal carotid artery. Thickness of the intima layer is measured at the middle third of the common carotid artery and is considered the measurement between the tunica intima and tunica media, the innermost two layers of the wall of an artery.
ophthalmic artery evaluation | 3-6 years after index pregnancy
  The woman is placed in a supine position to rest for 5 minutes. A 7.5-MHz linear transducer is then placed transversely and gently over her closed upper eyelid after application of conduction gel. Color flow Doppler is used to identify the ophthalmic artery, which is found superior and medially to the hypoechoic band representing the optic nerve. Pulsed-wave Doppler is then used to record 3 to 5 similar waveforms. Doppler studies are performed twice in each eye, and the average of the 4 measurements is used for analysis.
Cardiovascular markers in maternal blood | 3-6 years after index pregnancy
  Venous blood samples will be collected without anticoagulant to obtain serum. Placental growth factor (PlGF) will be measured in pg/ml using automated electrochemiluminescence immunoassays on the Roche Cobas platform (Roche Diagnostics GmbH, Mannheim, Germany).Intra-and interassay coefficients of variation were found to be <5%.
Laboratory data measured in g/l | 3-6 years after index pregnancy
  Venous blood samples and urine samples will be collected to measure hemoglobin and protein in urine
Laboratory data measured in l/l | 3-6 years after index pregnancy
  Venous blood samples will be collected to measure hematocrit
Laboratory data measured in U/mcl | 3-6 years after index pregnancy
  Venous blood samples will be collected to measure leukocytes and platalets
Laboratory data measured in mmol/l | 3-6 years after index pregnancy
  Venous blood samples will be collected to measure potassium and sodium
Laboratory data measured in % | 3-6 years after index pregnancy
  Venous blood samples will be collected to measure glicated hemoglobin
Laboratory data measured in U/L | 3-6 years after index pregnancy
  Venous blood samples will be collected to measure alanine transaminases, aspartate aminotransferases and lactate dehydrogenase
Laboratory data measured in mg/l | 3-6 years after index pregnancy
  Urine samples will be collected to measure albumin
Laboratory data measured in mUI/l | 3-6 years after index pregnancy
  Venous blood samples will be collected to measure tirotropin and prolactin
Ethnicity | 3-6 years after index pregnancy
  Patient ethnicity
Smoking status | 3-6 years after index pregnancy
  Patient smoking status
Menstrual type | 3-6 years after index pregnancy
  Patient menstrual type and presence of menopause
Diseases | 3-6 years after index pregnancy
  Diabetes, obesity, and other maternal diseases associated with cardiovascular risk
Interval from index preganancy | 3-6 years after index pregnancy
  interval in years from index pregnancy.
Gestational age at delivery | 3-6 years after index pregnancy
  Gestational age at delivery in index pregnancy
Mode of delivery | 3-6 years after index pregnancy
  mode of delivery at index pregnancy,
Labor induction | 3-6 years after index pregnancy
  labor induction at index pregnancy
Child's gender | 3-6 years after index pregnancy
  Child's gender in index pregnancy
Birth weight percentile | 3-6 years after index pregnancy
  birth weight percentile in index pregnancy
Birth weight | 3-6 years after index pregnancy
  Child's birth weight at index pregancy.
APGAR score | 3-6 years after index pregnancy
  5-minute Apgar score in index pregnancy. Apgar score measures appareance, pulse, grimance, acivity and respiratory effort. For each chriteria newborns can receive a punctuation from 0 to 2, qhere 2 is the better punctuation.
Blood preassure during pregnancy | 3-6 years after index pregnancy
  Blood preassure druing index pregnancy
Weight during pregnancy | 3-6 years after index pregnancy
  Weight during index pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Llurba, PhD, Principal Investigator — Hospital de la Sant Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i de Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brotons C, Moral I, Fernandez D, Puig M, Calvo Bonacho E, Martinez Munoz P, Catalina Romero C, Quevedo Aguado LJ. Estimation of Lifetime Risk of Cardiovascular Disease (IBERLIFERISK): A New Tool for Cardiovascular Disease Prevention in Primary Care. Rev Esp Cardiol (Engl Ed). 2019 Jul;72(7):562-568. doi: 10.1016/j.rec.2018.05.028. Epub 2018 Aug 7. English, Spanish. PMID 30097396
- [Background] Ferencik M, Pencina KM, Liu T, Ghemigian K, Baltrusaitis K, Massaro JM, D'Agostino RB Sr, O'Donnell CJ, Hoffmann U. Coronary Artery Calcium Distribution Is an Independent Predictor of Incident Major Coronary Heart Disease Events: Results From the Framingham Heart Study. Circ Cardiovasc Imaging. 2017 Oct;10(10):e006592. doi: 10.1161/CIRCIMAGING.117.006592. PMID 28956774
- [Background] Saenger AK, Beyrau R, Braun S, Cooray R, Dolci A, Freidank H, Giannitsis E, Gustafson S, Handy B, Katus H, Melanson SE, Panteghini M, Venge P, Zorn M, Jarolim P, Bruton D, Jarausch J, Jaffe AS. Multicenter analytical evaluation of a high-sensitivity troponin T assay. Clin Chim Acta. 2011 Apr 11;412(9-10):748-54. doi: 10.1016/j.cca.2010.12.034. Epub 2011 Jan 8. PMID 21219893
- [Background] Januzzi JL, van Kimmenade R, Lainchbury J, Bayes-Genis A, Ordonez-Llanos J, Santalo-Bel M, Pinto YM, Richards M. NT-proBNP testing for diagnosis and short-term prognosis in acute destabilized heart failure: an international pooled analysis of 1256 patients: the International Collaborative of NT-proBNP Study. Eur Heart J. 2006 Feb;27(3):330-7. doi: 10.1093/eurheartj/ehi631. Epub 2005 Nov 17. PMID 16293638
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2018 May 15;71(19):e127-e248. doi: 10.1016/j.jacc.2017.11.006. Epub 2017 Nov 13. No abstract available. PMID 29146535
- See also: IBERLIFERISK score — https://www.iberliferisk.com
- See also: REGICOR questionnaire — https://regicor.cat/en/applications/diet/
- See also: Phisycal activity questionnaire — https://regicor.cat/en/applications/physical-activity/